CLINICAL TRIAL: NCT07358351
Title: Feasibility of Robotic Instrument Guidance System to Perform Safe Ultrasound-Guided Percutaneous Procedures
Brief Title: Feasibility of Robotic Instrument Guidance System to Perform Safe Ultrasound-Guided Percutaneous Procedures During Routine Medical Procedures.
Acronym: ACCESS
Status: Active, not recruiting | Type: Observational
Sponsor: Mendaera, Inc (Industry)
Collaborators: CBCC Global Research LLP (Unknown)
Responsible Party: Sponsor
Other Study IDs: 100-00012-PROTOCOL-01
Record Dates: First submitted 2025-12-26; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Percutaneous Access
Keywords: ultrasound guided percutaneous access

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Prospective, single-center, single-arm: single arm
  Interventions: Device: Mendaera Guidance System

INTERVENTIONS:
Device: Mendaera Guidance System — Precise instrument placement of common percutaneous access devices for participants undergoing an ultrasound-guided procedure. Placement is conducted during routine care where percutaneous access is required.
  Other Names: Ultrasound guidance system

SUMMARY:
The Mendaera Guidance System ("Study Device") is intended to provide guidance for precise instrument placement of common percutaneous devices by positioning the device relative to the ultrasound transducer and the resulting image during a diagnostic or therapeutic procedure. After instrument placement is achieved, investigator will perform any further clinical tasks, procedures, or treatment using standard of care.

The target population for whom this device is intended includes participants requiring ultrasound guided, percutaneous procedures.

Participants who are scheduled to undergo an ultrasound-guided procedure will be consented and enrolled in the study.

Prior to the study procedure, participants should be prepared for ultrasound-guided procedure using standard of care.

Once the investigator determines that an ultrasound-guided procedure can be performed, the compatible percutaneous instrument will be connected to the Study Device, and the investigator may proceed to utilize the System to perform targeting and depth tracking of the instrument. Once access has been achieved, Participation will conclude after the first follow-up which is anticipated to be within 24±12 hours.

ELIGIBILITY:
Inclusion Criteria:

For all procedures:

* Age ≥ 18 years
* Subject or legal representative is willing and able to provide informed consent
* Subject is willing and able to comply with protocol follow-up
* Elective procedure (non-emergent)

For organ access procedures, one of the following must apply:

* Subjects for whom a percutaneous renal access for nephrostomy tube placement or percutaneous nephrolithotomy have has been indicated
* Subjects for whom a percutaneous biopsy have has been indicated
* Subjects for whom a percutaneous drainage (e.g. paracentesis, thoracentesis, etc.) have has been indicated

For vascular access procedures:

• Subjects for whom a vascular access (arterial or venous) have been indicated

For pain management injections procedures:

• Subjects for whom a pain management injection procedure has been indicated, such as intra-articular injection, nerve block pre- or post- operatively, and epidural

Exclusion Criteria:

* For all procedures:

  * Subject refusal
  * Subject is unstable or potentially unstable
  * Known significant coagulopathy (INR >2.0, platelet count <100,000 / µL)
  * Previous failed attempt of same procedure
  * Suspected infection at intended needle insertion or target site
  * BMI >35 kg/m²
  * Subject has any other medical, social, or psychological problem that, in the opinion of the Investigator, precludes them from participating
  * Subject who is pregnant or intends to become pregnant during the study
  * Hypertension (subject blood pressure ≥180/110mmHg)
  * History of venous thrombosis

For organ access procedures:

* Known anatomic abnormalities of target organ
* Subject underwent transplant or urinary diversion
* Abnormal kidney function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants undergoing an ultrasound-guided procedure
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2025-12-03 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Device-Related Adverse Events (occurrence and severity) | From enrollment to 24 hour follow-up (+/- 12 hours)
Number of participants with technical success defined as successful instrument placement using the device for the indicated procedure, as determined by the provider performing the procedure | Participant enrollment through 24 hour follow-up (+/- 12 hours)

SECONDARY OUTCOMES:
Time for relevant sub-steps of the procedure, including setup, draping, and access | Participant enrollment through 24 hour follow-up (+/- 12 hours)
Qualitative feedback and comparison of user's experience with the Mendaera system relative to standard of care | Participant enrollment through 24 hour follow-up (+/- 12 hours)
  User experience feedback on a scale of 1- to 5. How does the Mendaera system compare relative to standard of care?

CONTACTS AND LOCATIONS:
Locations (1):
- Mendaera, Inc, San Mateo, California, United States